CLINICAL TRIAL: NCT05666011
Title: A Single Center, Evaluator-Blinded, Split-Body, Randomized Pilot Study of Intense Pulsed Light Activation of Silver Nanoparticles vs. Intense Pulsed Light Alone in the Treatment of Keratosis Pilaris
Brief Title: Laser to Aid in Treatment of Keratosis Pilaris on Arms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KP-IPL
Record Dates: First submitted 2022-10-21; First posted 2022-12-27 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-10

CONDITIONS: Keratosis Pilaris
Keywords: keratosis pilaris; arms
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome; Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to combination treatment with IPL activation of SNA (i.e. intervention arm) versus IPL alone (i.e. control arm).
Who Masked: Investigator
Masking Description: Blinded Investigator will be unaware of which arm received which treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A -- Right side is Intervention Arm, Left side is Control Arm (Experimental): Right Arm will be treated with IPL activation of SNA (Silver Nanoparticles ) and left arm with IPL alone.
  Interventions: Device: M22 IPL
- Group B -- Left side is Intervention Arm, Right side is Control Arm (Experimental): Left Arm will be treated with IPL activation of SNA (Silver Nanoparticles ) and right arm with IPL alone.
  Interventions: Device: M22 IPL

INTERVENTIONS:
Device: M22 IPL — IPL is an attractive option in the treatment of KP as the provider can utilize cut-off filters to target both melanin for hair removal and erythema with a single device. An added benefit of IPL is the larger crystal size, allowing for efficient coverage of a larger body surface area. IPL has been utilized in the treatment of KP and KP variants, with outcomes showing reductions in both erythema and texture.
  Other Names: StellarM22 Intense Pulsed Light Laser

SUMMARY:
To assess efficacy and safety of intense pulsed light (IPL) activation of silver nanoparticles (SNA) versus IPL alone for treatment of keratosis pilaris.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess efficacy and safety of intense pulsed light (IPL; StellarM22™ Universal IPL, Lumenis Ltd., Yokneam, Israel) alone versus combination of IPL activation of silver nanoparticles (SNA) for treatment of keratosis pilaris.

Prior to first treatment, right and left arms of 10 enrolled subjects will be randomized to combination treatment with IPL activation of SNA (i.e. intervention arm) versus IPL alone (i.e. control arm). The intervention arm will be pre-treated with sugaring to epilate existing hair. This arm will then be treated with 0.5mL of nanoparticle suspension administered with a standard infusion paddle for 5 minutes prior to IPL treatment.

Following nanoparticle infusion, excess suspension will be removed from the surface of the skin with a pre-moistened wipe. Once all visible suspension is removed from the skin, the area will be cleansed with an alcohol wipe. If the alcohol wipe shows that the suspension is still present on the surface of the skin, additional pre-moistened wipes will be used to cleanse the skin until the alcohol wipe comes away without visible suspension. IPL will then be applied to the intervention arm.

Treatments will be repeated three times, spaced four- to six-weeks apart. After completing all three treatments, patients will return for macroscopic and dermoscopic photography at 1 month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 or older with clinical diagnosis of KP of the posterior upper arms.
* Subjects in good general health based on investigator's judgment and medical history
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study
* Understands and accepts the obligation and is logistically able to be present for all visits
* Is willing to comply with all requirements of the study and sign the informed consent documents
* Must be willing to maintain usual sun exposure for the duration of the study
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Subject agrees to avoid any changes in current skincare regimen.
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.

Exclusion Criteria:

* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* The subject is hypersensitive to light in the visible and/or near infrared wavelength region
* The subject is taking medication which is known to increase sensitivity to sunlight
* The subject has a seizure disorder triggered by light
* The subject has a pacemaker
* The subject has a metal implant that interferes with the transmission of energy to the electrical field
* The subject has any embedded electronic devices that give or receive a signal such as Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant
* Gold or metal allergy
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area or a neuropathic disorder
* The subject has used topical keratolytics, retinoids, chemical or mechanical exfoliative treatments in the 30 days prior to application of study treatment
* Dermal fillers, biostimulators, laser treatments, or other energy-based light treatments during the 6-month period before study treatment
* Subjects with tattoos in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, neoplasm of uncertain behavior, or untreated keratinocyte carcinoma/melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Erythema Grading Scale by a blinded investigator to assess change (one for each arm) | Baseline, Day 30, Day 60, Day 90, Day 110
  Erythema grading scale (Right Arm) 0 No erythema
  1. Mild erythema
  2. Moderate erythema
  3. Severe erythema
  4. Very severe erythema
  Erythema grading scale (Left Arm) 0 No erythema
  1. Mild erythema
  2. Moderate erythema
  3. Severe erythema
  4. Very severe erythema
Textural Change Grading Scale by a blinded investigator (one for each arm) | Baseline, Day 30, Day 60, Day 90, Day 110
  Textural change grading scale ( Right Arm) 0 No textural change
  1. Mild textural change
  2. Moderate textural change
  3. Severe textural change
  4. Very severe textural change
  Textural change grading scale (Left Arm) 0 No textural change
  1. Mild textural change
  2. Moderate textural change
  3. Severe textural change
  4. Very severe textural change
Investigator Global Aesthetic Improvement Scale (IGAIS) by a blinded investigator | Day 30, Day 60, Day 90, Day 110
  Blinded Physician Global Aesthetic Improvement Scale
  Rating Description
  1. Very Much Improved- Optimal cosmetic result in this subject
  2. Much Improved- Marked improvement in appearance form the initial condition, but not completely optimal for this subject.
  3. Improved- Obvious improvement in appearance from initial condition, but a re- treatment is indicated.
  4. No Change- The appearance is essentially the same as the original condition.
  5. Worse- The appearance is worse than the original condition.
  Scores (write a number under each treated area or check "Not Treated") Right Arm Left Arm
  Not Treated Not Treated

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (SGAIS) | Day 30, Day 60, Day 90, Day 110
  Subject Global Aesthetic Improvement Scale Assessment How would you rate the overall change in appearance of your treated areas? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description
  1. Very Much Improved- Optimal cosmetic result in this subject
  2. Much Improved- Marked improvement in appearance form the initial condition, but not completely optimal for this subject.
  3. Improved- Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change- The appearance is essentially the same as the original condition.
  5. Worse- The appearance is worse than the original condition.
  Scores (write a number under each treated area or check "Not Treated") Right Arm Left Arm
  Not Treated Not Treated

IPD SHARING:
Plan to Share IPD: Undecided